CLINICAL TRIAL: NCT05561101
Title: Evolution of the Health Status of Caregivers After the Admission of Their Elderly Relative to the Emergency Department
Acronym: ETAP-U
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A01294-39
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Caregiver-patient Dyeds; Patient Without Cognitive Disorders
Keywords: Caregiver-patient dyeds; Emergency Department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Caregivers burden — Assessment of caregiver burden after admision at Emergency Department of their elderly relative

SUMMARY:
The main objective of this non-interventional, propective and multipercentric study is to Assess the evolution of caregiver burden 1 month after their elderly relative's Emergency Department (ED) admission

DETAILED DESCRIPTION:
The aim purpose of this non-interventional, prospertive study is to compare the evolution of caregiver burden between inclusion and 1month after their elderly relative's ED admission.

Inclusion of caregivers - patients dyads, meeting inclusion criteria and agreeing to participate, is carried out by geriatric mobile teams (EMG) working within Emergengy Department.

At inclusion the following data will be collected:

For the patient :

* Presence of neurocognitive disorders
* Sociodemographic data (age, gender, lifestyle)
* Patient comorbidities
* Autonomy and independence
* Risk of early readmission and loss of autonomy

For the caregiver:

* Socio-demographic data
* The caregiver's burden
* Quality of life
* Resilience capacity will be measured

The follow-up of the caregiver is carried out 1 month after the passage of his elderly relative to Emergency Department (at inclusion). The levels of burden and quality of life as well as the aids set up at home will be collected

ELIGIBILITY:
Inclusion Criteria:

* Adult caregivers - patients aged 75 and over dyads consulting in Emergency Department and living at home
* Patients admitted to the emergency department for less than 48 hours for which a return home is decided
* Non-verbal opposition of the patient and caregiver to the collection of their data.

Exclusion Criteria:

* Hospitalized patient after emergency
* Patient admitted to emergency for life-saving emergency
* Patient living Nursing Home (EHPAD)
* Language barrier
* Absence of identified caregivers
* Severe cognitive impairment as per Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria and absence relative at time of inclusion
* Patients under guardianship
* Oral opposition from the patient and caregiver to their data collection.

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients - caregivers dyads aged 75 years and over, after admission to the elderly Emergency Department, without indication for hospitalization and living at home outside Nursing Home (EHPAD)
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-03-20 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
Measure of caregiver burden by the 7-item Zarit burden scale (Mini-zarit) | 1 month

SECONDARY OUTCOMES:
Assessment of patient's level of dependence through an appreciation of instrumental activities of daily living according Lawton scale | At inclusion
Assessment of the degree of patient dependence according "Index of Independence in Activities of Daily Living" KATZ scale | At inclusion
Assessment of complications risks according Triage Risk Screening Tool score (TRST) | At inclusion
Assessment of cognitive state of elderly patients according Abbreviated Mental Test 4 score (AMT-4) | At inclusion
  If score < 4 must search for neurocognitive disorders
Assessment of commorbidity risk according Charlson score | At inclusion
Assessment of quality of life of cargivers according SF-12 score | 1 month
Measure of caregiver satisfaction according Likert scale | 1 month
Measure of resilience capacities acoording Brief Resilience Scale (BRS) | At inclusion

CONTACTS AND LOCATIONS:
Overall Officials: PATRY Claire, MD, Study Chair — Extern Geriatric Mobile Team
Locations (1):
- Emergency Department, Bichat Hospital, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No